CLINICAL TRIAL: NCT03198403
Title: The Effect of Popliteal Plexus Block on Postoperative Pain After Total Knee Arthroplasty
Brief Title: The Effect of Popliteal Plexus Block on Pain After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Charlotte Runge, Consultant anesthetist, Principal investigator, Regionshospitalet Silkeborg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-001644-35
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Popliteal Plexus Block; Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Popliteal plexus block (Experimental): Patients with an FTB, reporting postoperative pain (NRS > 3) will have a popliteal plexus block
  Interventions: Drug: Bupivacaine-epinephrine
- No intervention (No Intervention): Patients with postoperative pain NRS < or = 3

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — Popliteal plexus block with 10 mL of bupivacaine-epinephrine 5 mg/mL + 5 microgram/mL.
  Arms: Popliteal plexus block

SUMMARY:
The study aims to investigate the effect of the Popliteal plexus block (PPB) on postoperative pain after total knee arthroplasty

DETAILED DESCRIPTION:
Cadaver dissection studies have shown a spread of dye to the popliteal fossa and colored the popliteal plexus by injecting in the distal part of the adductor Canal.

The popliteal plexus is formed by contribution from the tibial and the obturator nerves.

Investigators hypothesized that a PPB may reduce postoperative pain after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee arthroplasty in spinal anesthesia
* age > or = 18 years
* American Society of Anesthesiologists (ASA) status I-III
* Informed consent

Exclusion Criteria:

* Patients unable to cooperate
* Patients not able to speak Danish
* Pregnancy
* Contraindication towards ana Medical product used in the study
* Preoperatively reduced sensation on the medial and lateral part of the lower leg
* Patients with diabetic requiring Medical treatment
* Preoperative daily intake of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with postoperative pain NRS | 0 - 60 minutes
  Evaluated as the percentage of patients with postoperative pain NRS >3, dropping in pain score to NRS = or < 3 after the PPB

SECONDARY OUTCOMES:
Percentage of patients having a femoral triangle block(FTB) reporting NRS > 3 | Pain scores every 15 minutes (from end injection FTB to NRS>3 or 3 hours after full sensation of the leg)
  Percentage of patients having a FTB, reporting postoperative pain NRS >3
Onset time of PPB | NRS every 5 minutes after PPB (From 0 - 60 minutes after PPB)
  Time from end of injection of PPB to NRS = or < 3
Turn off time of spinal anesthesia | Time from arrival in PACU and during maximum 6 hours
  Time from arrival in PACU to normal cutaneous sensation (measured by a neuro-pen, sensation=point 2) on the lateral part of the thigh and lateral part of the lower leg
Correlation between normal cutaneous sensation and developing of pain | From arrival in PACU and during maximum 6 hours
  Correlation between normal cutaneous sensation (measured by a neuro-pen, sensation=point 2) and developing of pain (NRS>3)
The effect of the PPB on cutaneous sensation | NRS every 5 minutes after PPB (From 0 - 60 minutes after PPB)
  Tested on the lateral part of the lower leg
The effect of the PPB on muscle strength of the foot | Baseline and 1 hour after PPB
  Dorsal flexion and plantar flexion in the ankle joint, measured with a handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Runge, MD, Principal Investigator — University of Aarhus
Locations (1):
- Silkeborg Regionalhospital, Silkeborg, Denmark